CLINICAL TRIAL: NCT06862544
Title: Migraine Research with Smartwatch Application (MIRA) - a Prospective Migraine Study with Wearables
Brief Title: Migraine Research with Smartwatch Application
Acronym: MIRA
Status: Active, not recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: MIRA_1.0
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Migraine
Keywords: Migraine; Headache; Smartwatch; Wearables; Digital health tools
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Migraine patients: Patients with episodic or chronic migraine
  Interventions: Device: Smartwatch (Withings Scanwatch 2)

INTERVENTIONS:
Device: Smartwatch (Withings Scanwatch 2) — All-day monitoring of patients via smartwatch and migraine diary app

SUMMARY:
This clinical, prospective study aims to evaluate the effectiveness of wearable technology in capturing real-time data to assess disease activity in patients with episodic or chronic migraine undergoing different therapy strategies, including botulinum toxin, prophylactic, and acute treatments. Participants will also document migraine attacks, triggers, and symptoms through a digital migraine diary app. By combining continuous smartwatch data, the migraine diary and the implementation of questionnaires, the study seeks to provide a comprehensive understanding of how migraines and their treatments impact daily life and patient outcomes.

DETAILED DESCRIPTION:
Migraine is one of the most prevalent neurological disorders globally, significantly affecting patients' quality of life. However, due to the complexity of monitoring triggers and symptoms, determining the most effective individualized treatment regimen can be difficult. In this observational study a total of 55 patients with episodic or chronic migraines have been observed over a six-month period, with continuous data collection from both smartwatch and migraine diary app. Clinical health questionnaires were completed at baseline (V1), 3 months (V2), and 6 months (V3), assessing the impact of migraine attacks on daily functioning. The data gathered from the smartwatch (Withings ScanWatch) includes activity-related metrics (step count, minutes of activity at various intensity levels), basic cardiovascular measurements (heart rate), and sleep data (total sleep duration, sleep quality, etc.). Additionally, the Migraine App allows patients to document the precise timing of migraine attacks, associated symptoms, potential triggers, and the medications taken, including their effectiveness. The MIRA study aims to explore the potential of wearable devices and digital health tools to systematically identify migraine triggers and physiological responses through continuous monitoring. By integrating both clinical assessments and digital data, this study seeks to provide a comprehensive, longitudinal understanding of migraine dynamics and their impact on daily life.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be eligible to participate in the study:

* ≥ 18 years of age
* Diagnosed migraine syndrome
* Possession and ability to use a smartphone (Android 8.1 or later, or iOS 12.3 or later)

Exclusion Criteria:

* Missing informed consent
* Unwillingness or inability to use the smartphone app
* Comorbidity leading to impaired comprehension or successful completion of the study, such as (but not limited to) psychiatric comorbidities or dementia. The decision will be at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with episodic or chronic migraine 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
End-of-dose phenomena (EoD) in botulinum toxin therapy | Time Frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  The End-of-dose-phenomena-Questionnaire assesses the effectiveness of a treatment at the end of its dosing interval and asks about an increase in symptoms. Before their next botulinum toxin treatment, patients can state whether they have experienced a worsening of symptoms in recent weeks and, if so, for how many days and which migraine symptoms have worsened.
Change in Quality of life (QoL) | Time Frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  WHOQoL-BREF (World Health Organization Quality of Life Questionnaire Brief Version) is an instrument for measuring patients' subjective quality of life in a wide range of specific areas including Physical health, Psychological well-being, Social relationships and Environment. The WHOQoL-BREF uses a score range of 4 to 20 for each domain in its raw form. These raw scores are then converted to a 0-100 scale, where higher scores indicate better quality of life and lower scores indicate poorer quality of life.
Change in Migraine Disability (MIDAS) | Time Frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  MIDAS (Migraine Disability Assessment) is a standardized tool used to assess the impact of migraine on various aspects of life, including work, school, social activities, and leisure activities. It is calculated based on the number of days affected by migraines in the past three months with higher scores indicating greater disability and a more severe impact on daily activities. Lower scores suggest less disruption from migraines.
Change in Pittsburgh Sleep Quality Index (PSQI) | Time Frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  The Change in Pittsburgh Sleep Quality Index (PSQI) is a tool to assess the quality of sleep over the past month. The score range for the PSQI is from 0 to 21, with higher scores indicating poorer sleep quality.
Change in fatigue severity (BFI) | Time frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  Brief Fatigue Inventory (BFI) is a questionnaire to assess fatigue severity. The BFI consists of 9 questions, each answered on an 11-point scale. The total score on the BFI ranges from 0 to 10, where 0 represents no fatigue and 10 represents the worst possible fatigue. In general, higher scores indicate greater severity of fatigue, and lower scores suggest less severe or no fatigue.
Change in Depressive symptoms (BDI-FAST) | Time Frame: Screening + Baseline (V1), After 3 months (V2), After 6 months (V3)
  Beck Depression Inventory (BDI) FAST is a questionnaire to screen for depression in migraine patients. It is a shortened version of the full Beck Depression Inventory (BDI) and contains 7 items. Each item is scored on a 4-point scale (0 to 3), with a higher score indicating more severe depressive symptoms.
Smartwatch usage | After 6 months (V3)
  Questionnaire about smartwatch usage. Patients are presented with 17 statements about the smartwatches, focusing on practicality, usability, and everyday suitability. They can score each statement from 1 to 5, where 5 means strong agreement and 1 means strong disagreement.
Migraine Triggers | 180 days
  Migraine Triggers through migraine diary
Medication taken during migraine attacks | 180 days
  Medication taken during migraine attacks through migraine diary
Duration of migraine attacks | 180 days
  Duration of migraine attacks through migraine diary
Pain level and localization of headache | 180 days
  Pain level and localization of headache through migraine diary. For each migraine attack there is a Numerical Rating Scale (NRS) - a simple method for pain assessment, where patients rate their pain on a scale from 0 to 10. In the migraine app, patients can specify the exact location of their headache. A front view of the head with 12 sections and a back view with 6 sections are presented. Patients can select multiple sections to visually pinpoint the headache location.
Wearing time of smartwatch (daily) | 180 days
Longitudinal development of activity parameter: step count | 180 days
Longitudinal development of activity parameter: approximate distance traveled (meter) | 180 days
Longitudinal development of activity parameter: duration of soft activity (seconds) defined by Withings Description: Examples for soft activity: Sleeping, Sitting quietly, Walking slowly, Typing on a computer keyboard while seated, Watching televisio | 180 days
Longitudinal development of activity parameter: duration of moderate activity (seconds) defined by Withings Description: Examples for moderate activity: Walking fast, Cleaning (vacuuming, washing windows, etc.), Playing doubles tennis or badminton, T | 180 days
Longitudinal development of activity parameter: duration of intense activity (seconds) defined by Withings Description: Examples for intense activity: Hiking, Running, Carrying heavy loads, Riding a bike, Playing football, baseball, or tennis (singles), | 180 days
Longitudinal development of activity parameter: sum of all active time (seconds) | 180 days
Longitudinal development of activity parameter: approximate calories burned Time | 180 days
Longitudinal development of sleep parameter: time awake (seconds) | 180 days
Longitudinal development of sleep parameter: number of times user woke up | 180 days
Longitudinal development of sleep parameter: time to sleep (seconds) | 180 days
Longitudinal development of sleep parameter: total time in bed (seconds) | 180 days
Longitudinal development of sleep parameter: total time asleep (seconds) | 180 days
Longitudinal development of sleep parameter: ratio of sleep/time in bed | 180 days
Longitudinal development of sleep parameter: time spent in bed before falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: time awake after first falling asleep (seconds) | 180 days
Longitudinal development of sleep parameter: Withings Sleep score Description: Defined by Withings as follows: It measures every night's sleep and provides a score out of 100 points based on 4 key inputs: - Duration (total time spent sleeping) - Depth (p | 180 days
Longitudinal development of cardiovascular parameter: average heartrate | 180 days
Longitudinal development of cardiovascular parameter: maximal heartrate | 180 days
Longitudinal development of cardiovascular parameter: minimum heartrate | 180 days
Longitudinal development of cardiovascular parameter: time in light heartrate zone (seconds) Description: Light heartrate zone is defined by Withings as follows: from 0% inclusive to 50% exclusive of maximum heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in moderate heartrate zone (seconds) Description: Moderate heartrate zone is defined by Withings as follows: from 50% included to 70% excluded of maximal heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in intense heartrate zone (seconds) Description: Intense heartrate zone is defined by Withings as follows: from 70% included to 90% excluded of maximal heart rate. | 180 days
Longitudinal development of cardiovascular parameter: time in maximal heartrate zone (seconds) Description: Maximal heartrate zone is defined by Withings as follows: from 90% included to 100% included of maximal heart rate | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty, Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No